CLINICAL TRIAL: NCT05457387
Title: Examining the Association Between Perioperative Sleep Disturbance and Postoperative Delirium During Non-cardiac Surgery
Brief Title: Relationship Between Perioperative Sleep Disturbance and Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Fudan University (Other); Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Taihe Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-POD-002
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are performing this research study to understand the role of sleep disturbance on the incidence of delirium after surgery.

DETAILED DESCRIPTION:
Sleep is one of the most important physiological needs. Sleep disturbances have detri-mental effects on practically all systems and may thus prolong recovery of patients. Studies have documented many similarities between clinical and physiological profiles of patients with delirium and sleep disturbances (ischemia/inflammation, hypoxia, neu-rotransmitter imbalance and tryptophan/melatonin metabolism abnormalities). There is still a lack of strong evidence to support the link between poor sleep and delirium, par-ticularly in hospitalized patients, even though available studies suggest that sleep dis-turbances may be a potential key risk factor for its development, which may have a significant clinical impact.

Post operative delirium will be diagnosed using the 3D- CAM(Confusion Assessment Method) which tests for four features with a series of questions. The features include 1) acute onset and fluctuating course,2) inattention,3) disorganized thinking and 4) altered level of consciousness. Diagnosis of delirium is made if features 1 and 2 and either 3 or 4 are present.

The demographic data of the patients,type and site of surgery will be noted. Preoperative hemoglobin, serum electrolytes and blood urea will be recorded. The intraoperative factors like duration of surgery and anaesthesia,use of intravenous fluids ,blood loss, number blood units transfused and opioid use will be studied at the time of surgery. The time to emergence and extubation following the completion of surgery will be noted.

The association of various preoperative,intraoperative and postoperative factors with POD will be determined.

ELIGIBILITY:
Inclusion Criteria:

Geriatric surgical patients ≥65 years old

Exclusion Criteria:

Patients in the central nervous system group were excluded from cardiac and neurosurgery, patients in the heart injury group were excluded from cardiac surgery, and patients who did not agree to participate in the study were excluded in all groups.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 11927 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 7 days post surgery
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
the incidence of survival rate | 1 year
  collection of clinical data in the medical record and follow-up update
Sleep NRS | 1 day before the surgery
  sleep numerical rating scale
Sleep NRS | 7 days post surgery
  sleep numerical rating scale
Sleep NRS | baseline
  sleep numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Weidong G Mi, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided